CLINICAL TRIAL: NCT04917536
Title: Comparison Between the Entry Portals Through the Rotator Cuff and Through the Rotator Interval Split for Anterograde Humeral Nailing in Humeral Fractures: a Prospective Randomized Study
Brief Title: Comparison of the Speed of Functional Recovery (Constant Score) Between Two Different Approaches of Humeral Nailing in Humeral Fractures: Through the Rotator Cuff or Through the Rotator Interval Split (HUNAAP)
Acronym: HUNAAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2021 VILLATTE; 2021-A00400-41 (Other: ANSM)
Record Dates: First submitted 2021-05-20; First posted 2021-06-08 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Humeral Upper Extremity Fracture; Humeral Diaphysis Fracture
Keywords: Speed of functional recovery; Humeral fractures; Anterograde nailing; Rotator cuff split; Prospective randomized study
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Intervention Model Description: Approach through the rotator cuff or through the rotator cuff split
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rotator cuff approach (Active Comparator): the nail is inserted through the supra-spinatus tendon, which is closed at the end of the surgery
  Interventions: Procedure: Humeral neailling in humeral fractures
- rotator cuff split approach (Experimental): the nail is inserted through the rotator cuff split, between the supra-spinatus tendon and the long part of the biceps
  Interventions: Procedure: Humeral neailling in humeral fractures

INTERVENTIONS:
Procedure: Humeral neailling in humeral fractures — Humeral neailling in humeral fractures

SUMMARY:
The aim of the study is to show if there is any speed difference of functional recovery for people with humeral fracture, treated by an anterograde nail, which will be inserted through the rotator cuff (the common way) or through the rotator interval split.

The patients included in this study will be randomized to one of the two groups.

The recovery will be evaluated by the Constant score over time, for a year. The main hypothesis is the rotator interval split approach allows a faster functional recovery after humeral nailing, by avoiding opening the rotator cuff.

DETAILED DESCRIPTION:
Humeral fractures are the third most common fractures over 65 years and represent 8% of all fractures. The anterograde nailing is known to be an efficient way to treat humeral upper extremity fractures and humeral diaphysis fractures. The main complications of this nailing are pain, shoulder stiffness, rotator cuff tendinitis and impingement.

Studies have proven these problems can be due to the entry portal of the nail. Indeed, it is inserted through the supra-spinatus tendon, which means an opening of the rotator cuff even if it is closed at the end of the procedure.

But the rotator interval split in the shoulder can allow to insert the nail through it without opening the cuff or damaging the cartilage. It is located between the anterior side of the supra-spinatus tendon and the posterior side of the long part of the biceps.

The aim of the study is to compare the speed of functional recovery according to the entry portal, which are through the rotator cuff or through the rotator interval split, in humeral fractures treated by anterograde nailing.

The cutaneo-muscular approach will be the same in both groups, namely a trans-deltoid approach.

People will be included in the study after an enlightened and signed consent, afterward they will be randomized to one of the two groups.

To evaluate the primary outcome, the Constant Score will be used to measure the kinetic of the recovery.

The secondary outcomes are residual pain (measured by the VAS an evaluation of complications and a radiological review (two different reviewers) to follow the healing and search any side effects, the sick leave and rehabilitation durations.

The patients need to be available for a one-year follow-up. Each assessment will be checked at 21 and 45 days, and at 3, 6 and 12 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Be available for a one year follow-up
* Patients over 18 and under 70 years old
* Humeral diaphysis fracture or humeral upper extremity articular fracture (Neer 2,3 or 4), needing to be treated by anterograde nailing.
* No growth plates
* Patients covered by the French social security service
* Patients able to give their enlightened consent and to answer the questions asked for the trial

Exclusion Criteria:

* Pregmant, breastfeeding or potentially pregmant woman
* Existing bone disease
* Polytrauma
* Other fractures on the same upper limb
* Pathologic fracture
* Medical history of surgery on the same shoulder
* Contra-indication to the surgery or the anesthesia
* Infection on the operating site
* Axillary nerve palsy
* Deltoid dysfunction
* Major disability
* Refusal of participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Speed of functional recovery | Day 21
  Measured by the objective Constant score (absolute and weighted values), which includes an evaluation of the pain, level of daily activities, use of the hand, range of motion and strength. The collected data will allow us to draw a diagram to compare the speed of recovery. Its values are between 0 (bad) and 100 (good)
Speed of functional recovery | Day 45
  Measured by the objective Constant score (absolute and weighted values), which includes an evaluation of the pain, level of daily activities, use of the hand, range of motion and strength. The collected data will allow us to draw a diagram to compare the speed of recovery. Its values are between 0 (bad) and 100 (good)
Speed of functional recovery | Month 3
  Measured by the objective Constant score (absolute and weighted values), which includes an evaluation of the pain, level of daily activities, use of the hand, range of motion and strength. The collected data will allow us to draw a diagram to compare the speed of recovery. Its values are between 0 (bad) and 100 (good)
Speed of functional recovery | Month 6
  Measured by the objective Constant score (absolute and weighted values), which includes an evaluation of the pain, level of daily activities, use of the hand, range of motion and strength. The collected data will allow us to draw a diagram to compare the speed of recovery. Its values are between 0 (bad) and 100 (good)
Speed of functional recovery | Month 12
  Measured by the objective Constant score (absolute and weighted values), which includes an evaluation of the pain, level of daily activities, use of the hand, range of motion and strength. The collected data will allow us to draw a diagram to compare the speed of recovery. Its values are between 0 (bad) and 100 (good)

SECONDARY OUTCOMES:
Quick Dash | Day 21
  subjective test showing any difficulties in the daily living activities, relationships, and evaluating the pain and tingling; all of these items are based on the week before the assessment. It ranges from 0 to 100 more the value is better brought up is the score.
Quick Dash | Day 45
  subjective test showing any difficulties in the daily living activities, relationships, and evaluating the pain and tingling; all of these items are based on the week before the assessment. It ranges from 0 to 100 more the value is better brought up is the score.
Quick Dash | Month 3
  subjective test showing any difficulties in the daily living activities, relationships, and evaluating the pain and tingling; all of these items are based on the week before the assessment. It ranges from 0 to 100 more the value is better brought up is the score.
Quick Dash | Month 6
  subjective test showing any difficulties in the daily living activities, relationships, and evaluating the pain and tingling; all of these items are based on the week before the assessment. It ranges from 0 to 100 more the value is better brought up is the score.
Quick Dash | Month 12
  subjective test showing any difficulties in the daily living activities, relationships, and evaluating the pain and tingling; all of these items are based on the week before the assessment. It ranges from 0 to 100 more the value is better brought up is the score.
Simple shoulder test (SST) | day 21
  a subjective score to evaluate what kind of activity is actually possible for the patient
Simple shoulder test (SST) | day 45
  a subjective score to evaluate what kind of activity is actually possible for the patient
Simple shoulder test (SST) | Month 3
  a subjective score to evaluate what kind of activity is actually possible for the patient
Simple shoulder test (SST) | Month 6
  a subjective score to evaluate what kind of activity is actually possible for the patient
Simple shoulder test (SST) | Month 12
  a subjective score to evaluate what kind of activity is actually possible for the patient
Intensity of Pain | Day 21
  Visual analog scale (VAS) : the pain is quantified by a number from 0 (no pain) to 10 (the worst pain ever known)
Intensity of Pain | Day 45
  Visual analog scale (VAS) : the pain is quantified by a number from 0 (no pain) to 10 (the worst pain ever known)
Intensity of Pain | Month 3
  Visual analog scale (VAS) : the pain is quantified by a number from 0 (no pain) to 10 (the worst pain ever known)
Intensity of Pain | Month 6
  Visual analog scale (VAS) : the pain is quantified by a number from 0 (no pain) to 10 (the worst pain ever known)
Intensity of Pain | Month 12
  Visual analog scale (VAS) : the pain is quantified by a number from 0 (no pain) to 10 (the worst pain ever known)
Complications assessment | day 0
  Searching any early or late complications, such as neurological or vascular problems, haematoma, infection, dislocation, with a clinical exam or other possible paraclinical exams
Complications assessment | day 21
  Searching any early or late complications, such as neurological or vascular problems, haematoma, infection, dislocation, with a clinical exam or other possible paraclinical exams
Complications assessment | day 45
  Searching any early or late complications, such as neurological or vascular problems, haematoma, infection, dislocation, with a clinical exam or other possible paraclinical exams
Complications assessment | Month 3
  Searching any early or late complications, such as neurological or vascular problems, haematoma, infection, dislocation, with a clinical exam or other possible paraclinical exams
Complications assessment | Month 6
  Searching any early or late complications, such as neurological or vascular problems, haematoma, infection, dislocation, with a clinical exam or other possible paraclinical exams
Complications assessment | Month 12
  Searching any early or late complications, such as neurological or vascular problems, haematoma, infection, dislocation, with a clinical exam or other possible paraclinical exams
Duration of the sick leave | day 21
  The patient is asked when he has returned to his professional activity
Duration of the sick leave | day 45
  The patient is asked when he has returned to his professional activity
Duration of the sick leave | Month 3
  The patient is asked when he has returned to his professional activity
Duration of the sick leave | Month 6
  The patient is asked when he has returned to his professional activity
Duration of the sick leave | Month 12
  The patient is asked when he has returned to his professional activity
Duration of the rehabilitation | day 21
  The patient is asked about the length of the physiotherapy.
Duration of the rehabilitation | day 45
  The patient is asked about the length of the physiotherapy.
Duration of the rehabilitation | month 3
  The patient is asked about the length of the physiotherapy.
Duration of the rehabilitation | month 6
  The patient is asked about the length of the physiotherapy.
Duration of the rehabilitation | month 12
  The patient is asked about the length of the physiotherapy.
Surgery datas | during the surgery and immediately after (Day 0)
  any or no transfusion of blood cells
Surgery datas | during the surgery (Day 0)
  time to perform the surgery collected from the operating file in minutes
haemoglobin levels | during the surgery and immediately after (Day 0)
  haemoglobin levels in g/dl
Radiological evolution | Day 45
  consolidation or not
Radiological evolution | Month 3
  consolidation or not
Radiological evolution | Month 6
  consolidation or not
Radiological evolution | Month 12
  consolidation or not

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Villatte, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France